CLINICAL TRIAL: NCT05533905
Title: DECISIve - DiagnosE Using the Central veIn SIgn. A Prospective Diagnostic Superiority Study Comparing T2*MRI and Lumbar Puncture in Patients Presenting With Possible Multiple Sclerosis.
Brief Title: DECISIve - DiagnosE Using the Central veIn SIgn v1.0
Acronym: DECISiVE
Status: Completed | Type: Observational
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 19NS022
Record Dates: First submitted 2022-09-06; First posted 2022-09-09 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Spinal Puncture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Lumbar puncture — A thin needle is inserted between the bones in the spine.
Diagnostic Test: MRI — A scan of the head.

SUMMARY:
DECISIve - DiagnosE using the Central veIn SIgn. A prospective diagnostic superiority study comparing T2* MRI and lumbar puncture in patients presenting with possible Multiple Sclerosis

DETAILED DESCRIPTION:
There is currently no agreement on the best way to diagnose Multiple Sclerosis (MS). Frequently, people suspected of having MS have a standard MRI scan and undergo a 'lumbar puncture' (a thin needle is inserted between the bones in the lower spine). Patients often report they find it painful and it can cause unintended complications requiring hospitalisations or time off work to recover.

Although the fluid taken during a lumbar puncture can show evidence of disease, this is not always the case. We do not find abnormalities in everyone who has MS but some people with conditions that can mimic MS, but need very different treatment, have similar lumbar puncture abnormalities. Both of these problems can lead to misdiagnosis.

A new MRI scan allows us to see small veins that run through damaged areas of the brain in people with MS. It has been shown that this is a specific finding to MS, seldom seen in other conditions. It is not painful and carries few or no risks.

This research aims to change the way people are diagnosed with MS and reduce the number of lumbar punctures used. Our team will recruit a large number of people from different hospitals whose doctors suspect they may have MS. We will invite them to have the new eight-minute MRI scan. After 18 months, we will find out what diagnosis is eventually reached and compare this to the finding of the new scan. We will compare the accuracy, speed, costs and acceptability of the different tests needed to make a diagnosis of MS and establish if most lumbar punctures can be replaced by a slightly longer MRI scan. This research could provide the NHS with a scientific approach to diagnose MS which is safer, more cost effective and importantly, more acceptable to patients.

ELIGIBILITY:
Inclusion Criteria:

* Presentation with a typical clinically isolated syndrome (Thompson et al. 2017) for diagnostic evaluation of MS.

Exclusion Criteria:

1. Fulfils the diagnosis of MS, as defined by the 2017 revision of McDonald diagnostic criteria (Thompson et al. 2017).
2. Unwilling or unable to comply with the requirements of this protocol including the presence of any condition (physical, mental, or social) that, in the opinion of the PI, is likely to affect the participant's ability to comply with the study protocol.
3. Unable to provide informed consent.
4. Contraindication or inability to undergo MRI due to metal or metal implants, pregnancy, claustrophobia, pain, spasticity, or excessive movement related to tremor.
5. Acute COVID-19 infection at time of face-to-face interactions during study (unless investigations can be delayed until considered safe by the responsible clinician and PI) either diagnosed clinically or by acute infection testing
6. Participant required to self-isolate at time of face-to-face interactions during study (unless investigations can be delayed until considered safe by the responsible clinician and PI) due to COVID-19 exposure, shielding due to medical advice, public health advice or governmental advice/laws.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 115 participants will be recruited over 30 months across the four participating sites.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2023-11-06 (Actual); Study Completion 2023-11-06 (Actual)

PRIMARY OUTCOMES:
Is T2* MRI scan more sensitive than lumbar puncture with oligoclonal band testing for diagnosing MS at the time of first clinical presentation? | 18 months
  Comparison of MRI and lumbar puncture in diagnosing MS.

SECONDARY OUTCOMES:
Is there a significant difference between the specificity of each diagnostic test in this cohort? | 18 months
  Is there a difference in the quality of the diagnostic tests.
Is there a significant difference between the sensitivity and specificity of the 'rule of six' proposed in Mistry et al. 2016 and lumbar puncture with oligoclonal bands? | 18 months
  Comparison with past research

CONTACTS AND LOCATIONS:
Overall Officials: Nikos Evangelou, Principal Investigator — NUH NHS Trust
Locations (1):
- NUH NHS Trust, Nottingham, United Kingdom